CLINICAL TRIAL: NCT01998477
Title: A Phase III, Observer-Blind, Randomized Multicenter Study to Evaluate the Safety of Trivalent Subunit Influenza Vaccines, Produced Either in Mammalian Cell Culture (TIVc) or in Embryonated Eggs (TIV), in Children and Adolescents 3 to <18 Years of Age at Risk for Influenza-Related Complications
Brief Title: A Study to Evaluate the Safety of Two Influenza Vaccines in Children and Adolescents 3 to <18 Years of Age at Risk for Influenza-Related Complications
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V58P15; 2013-002080-26 (EudraCT Number)
Record Dates: First submitted 2013-10-30; First posted 2013-11-29 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Influenza
Keywords: Influenza; Vaccine; Flu; Children; Adolescents
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TIVc (Experimental): flu vaccine
  Interventions: Biological: TIVc
- TIV (Active Comparator): flu vaccine
  Interventions: Biological: TIV

INTERVENTIONS:
Biological: TIVc — Madin Darby Canine Kidney (MDCK) cell culture derived subunit influenza vaccine TIVc contained the purified viral envelope glycoproteins, hemagglutinin (HA) and neuraminidase (NA) derived from 3 strains (including HA for each strain [A/H1N1-like, A/H3N2-like, and B-like]) intramuscular (IM) injection recommended by the WHO for the 2013-2014 influenza season in the Northern Hemisphere
  Arms: TIVc
Biological: TIV — A conventional egg derived subunit influenza vaccine (TIV) contained the purified viral envelope-glycoproteins, HA and NA derived from 3 strains (including HA for each strain [A/ H1N1-like, A/H3N2-like, and B-like]) IM injection recommended by the WHO for the 2013-2014 influenza season in the Northern Hemisphere.
  Arms: TIV

SUMMARY:
The study is designed to evaluate the safety of TIVc or TIV vaccine in children 3 to < 18 years of age who are at risk of complications of influenza disease due to underlying diseases.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 3 to <18 years of age with underlying medical conditions that indicate an increased risk of complications from influenza infection.
* Further eligibility criteria may be discussed by contacting the site(s)

Exclusion Criteria:

* Individuals with any fatal prognosis of an underlying medical condition (<12 month life expectancy).
* Individuals hospitalized at the time of enrolment.
* Individuals with a history of any anaphylaxis, serious vaccine reactions, or hypersensitivity to any of the vaccine components.
* Further eligibility criteria may be discussed by contacting the site(s)

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 430 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (16):
- Italy (4):
  - Novartis Investigational Site 022, Florence
  - Novartis Investigational Site 020, Genova
  - Novartis Investigational Site 021, Milan
  - Novartis Investigational Site 023, Roma
- Spain (12):
  - Novartis Investigational Site 031, Badalona, Barcelona
  - Novartis Investigational Site 017, Burriana, Castellon
  - Novartis Investigational Site 016, Castellon, Castellon
  - Novartis Investigational Site 010, Marbella, Malaga
  - Novartis Investigational Site 015, L'Eliana, Valencia
  - Novartis Investigational Site 013, Paiporta, Valencia
  - Novartis Investigational Site 018, Quart de Poblet, Valencia
  - Novartis Investigational Site 030, Madrid
  - Novartis Investigational Site 011, Málaga
  - Novartis Investigational Site 019, Valencia
  - Novartis Investigational Site 014, Valencia
  - Novartis Investigational Site 012, Valencia

REFERENCES:
- [Derived] Diez-Domingo J, de Martino M, Lopez JG, Zuccotti GV, Icardi G, Villani A, Moreno-Perez D, Hernandez MM, Aldean JA, Mateen AA, Enweonye I, de Rooij R, Chandra R. Safety and tolerability of cell culture-derived and egg-derived trivalent influenza vaccines in 3 to <18-year-old children and adolescents at risk of influenza-related complications. Int J Infect Dis. 2016 Aug;49:171-8. doi: 10.1016/j.ijid.2016.06.018. Epub 2016 Jun 23. PMID 27343983

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 12 centers in Spain and 4 centers from Italy.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- TIVc (3 to <18 Years): Vaccine naive and non-naïve subjects received one or two doses of cell culture derived trivalent subunit influenza vaccine formulation (TIVc)
- TIV (3 to <18 Years): Vaccine naive and non-naïve subjects received one or two doses of egg derived trivalent subunit influenza vaccine formulation (TIV)
Period: Overall Study
Arm/Group | TIVc (3 to <18 Years) | TIV (3 to <18 Years)
Started | 282 | 148
Completed | 272 | 143
Not Completed | 10 | 5
Not completed — Lost to Follow-up | 4 | 5
Not completed — Withdrawal by Subject | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TIVc (3 to <18 Years) | TIV (3 to <18 Years) | Total
Number analyzed (Participants) | 282 | 148 | 430
Age, Continuous [Mean (Standard Deviation); unit: year] | 8.7 (4.0) | 9.0 (3.9) | 8.8 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  FEMALE | 121 | 63 | 184
  MALE | 161 | 85 | 246

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Solicited Adverse Events (AEs) Following Vaccination With Either TIVc or TIV by Overall Age Group
Description: Safety was assessed in terms of number of the subjects (3 to < 18 years of age) who reported solicited local, systemic AEs as well as other solicited AEs after receiving one or two doses of either TIVc or TIV
Time Frame: Day 1 through Day 7 post injection 1 and Day 29 through Day 35 post injection 2
Population: Analysis was done on safety dataset, i.e. the subjects in the Exposed Set who provided post-vaccination solicited AE data
Measure: Number; unit: Subjects
Groups:
- TIVc _inj 1 (3 to <18 Years); TIVc_inj 2 (3 to <18 Years): Vaccine naive and non-naïve subjects received one or two doses of cell culture derived trivalent subunit influenza vaccine formulation (TIVc)
- TIV_inj 1 (3 to <18 Years); TIV_inj 2 (3 to <18 Years): Vaccine naïve and non-naive subjects received one or two doses of egg derived trivalent subunit influenza vaccine formulation (TIV)
Arm/Group | TIVc _inj 1 (3 to <18 Years) | TIVc_inj 2 (3 to <18 Years) | TIV_inj 1 (3 to <18 Years) | TIV_inj 2 (3 to <18 Years)
Number analyzed (Participants) | 277 | 83 | 145 | 40
Subjects
  Any Local | 149 | 41 | 89 | 18
  Injection Site Tenderness | 25 | 20 | 17 | 6
  Injection Site Pain | 106 | 19 | 65 | 8
  Injection site erythema ,< 6 years | 8 | 3 | 4 | 4
  Injection site induration < 6 years | 7 | 5 | 4 | 3
  Injection site ecchymosis < 6 years | 6 | 1 | 3 | 3
  Injection site erythema >=6 years | 16 | 5 | 22 | 3
  Injection site induration >=6years | 22 | 3 | 23 | 3
  Injection site ecchymosis >= 6 years | 8 | 2 | 5 | 5
  Any Systemic | 117 | 29 | 55 | 8
  Change in eating habits | 12 | 6 | 7 | 2
  Chills | 32 | 6 | 9 | 0
  Diarrhea | 19 | 2 | 5 | 3
  Irritability | 14 | 5 | 7 | 2
  Sleepiness | 10 | 5 | 3 | 2
  Vomiting | 18 | 3 | 5 | 1
  Arthralgia | 24 | 0 | 9 | 0
  Fatigue | 28 | 4 | 16 | 0
  Headache | 35 | 8 | 24 | 1
  Loss of appetite | 30 | 5 | 16 | 2
  Myalgia | 35 | 5 | 14 | 0
  Nausea | 21 | 0 | 12 | 0
  Body Temp. ( >= 38C ) | 18 | 2 | 6 | 0
  Treatment of pain and or fever | 28 | 7 | 11 | 1
  Prevention of pain and or fever | 19 | 2 | 9 | 3

2. Primary Outcome: Number of Subjects Reporting Solicited Adverse Events (AEs), Following Vaccination With Either TIVc or TIV by Age Sub-strata
Description: Safety was assessed in terms of number of the subjects (3 to <6 years,(≥ 6 to < 9 years and 9 to <18 Years of age) who reported solicited local, systemic AEs as well as other solicited AEs after receiving one or two doses of either TIVc or TIV
Time Frame: Day 1 through Day 7 after any vaccination
Population: Analysis was done on safety dataset
Measure: Number; unit: Subjects
Groups:
- TIVc_Non naive_inj 1 (3 to <6 Years); TIVc_Non naive_Inj 1 (≥ 6 to < 9 Years): Vaccine non-naïve subjects received one dose of cell culture derived trivalent subunit influenza vaccine formulation (TIVc)
- TIVc_naive_inj 1 (3 to <6 Years); TIVc_naive_inj 2 (3 to <6 Years); TIVc_Naive_inj 1 (≥ 6 to < 9 Years); TIVc_Naive_inj 2 (≥ 6 to < 9 Years): Vaccine naïve subjects received two doses of cell culture derived trivalent subunit influenza vaccine formulation (TIVc)
- TIV_Non naive_inj 1 (3 to <6 Years); TIV_Non Naive (9 to <18 Years): Vaccine nonnaïve subjects received one dose of egg derived trivalent subunit influenza vaccine formulation (TIV)
- TIV_naive_inj 1 (3 to <6 Years); TIV_naive_inj 2 (3 to <6 Years); TIV_Naive_inj 1 (≥ 6 to < 9 Years); TIV_Naive_inj 2 (≥ 6 to < 9 Years): Vaccine naïve subjects received two doses of egg derived trivalent subunit influenza vaccine formulation (TIV)
- TIV_Non Naive_inj 1 (≥ 6 to < 9 Years): Vaccine non-naïve subjects received one dose of egg derived trivalent subunit influenza vaccine formulation (TIV)
- TIVc_Non Naive (9 to <18 Years): Vaccine nonnaïve subjects received one dose of cell culture derived trivalent subunit influenza vaccine formulation (TIVc)
Arm/Group | TIVc_Non naive_inj 1 (3 to <6 Years) | TIVc_naive_inj 1 (3 to <6 Years) | TIVc_naive_inj 2 (3 to <6 Years) | TIV_Non naive_inj 1 (3 to <6 Years) | TIV_naive_inj 1 (3 to <6 Years) | TIV_naive_inj 2 (3 to <6 Years) | TIVc_Non naive_Inj 1 (≥ 6 to < 9 Years) | TIVc_Naive_inj 1 (≥ 6 to < 9 Years) | TIVc_Naive_inj 2 (≥ 6 to < 9 Years) | TIV_Non Naive_inj 1 (≥ 6 to < 9 Years) | TIV_Naive_inj 1 (≥ 6 to < 9 Years) | TIV_Naive_inj 2 (≥ 6 to < 9 Years) | TIVc_Non Naive (9 to <18 Years) | TIV_Non Naive (9 to <18 Years)
Number analyzed (Participants) | 28 | 50 | 50 | 19 | 15 | 15 | 26 | 35 | 33 | 16 | 23 | 24 | 138 | 72
Subjects
  Any Local | 14 | 19 | 22 | 12 | 7 | 7 | 16 | 19 | 19 | 8 | 13 | 11 | 81 | 49
  Tenderness(N=28,49,49,19,15,15,0,0,0,0,0,0,0,0) | 10 | 15 | 20 | 11 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain(N=0,0,0,0,0,0,26,32,31,16,22,22,138,72) | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 18 | 19 | 8 | 10 | 8 | 73 | 47
  Erythema27,50,50,18,15,15,26,34,32,16,23,23,131,61 | 7 | 1 | 3 | 4 | 0 | 4 | 1 | 3 | 5 | 4 | 5 | 3 | 5 | 2
  Injection site induration | 2 | 5 | 5 | 2 | 2 | 3 | 1 | 4 | 3 | 3 | 2 | 3 | 6 | 7
  Injection site ecchymosis | 2 | 4 | 1 | 2 | 1 | 3 | 2 | 3 | 2 | 0 | 3 | 5 | 0 | 0
  Any Systemic | 10 | 22 | 14 | 9 | 5 | 5 | 9 | 18 | 15 | 5 | 5 | 3 | 58 | 31
  Change in eating habits | 5 | 7 | 6 | 3 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills28,50,48,19,15,14,25,33,31,16,22,23,138,72 | 2 | 5 | 3 | 2 | 0 | 0 | 3 | 3 | 3 | 1 | 0 | 0 | 19 | 6
  Diarrhea28,50,50,19,14,15,26,33,31,16,22,23,137,71 | 3 | 1 | 1 | 1 | 0 | 2 | 1 | 3 | 1 | 0 | 0 | 1 | 11 | 4
  Irritability | 6 | 8 | 5 | 5 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sleepiness(N=28,49,48,19,15,15,0,0,0,0,0,0,0,0) | 4 | 6 | 5 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Vomiting28,50,50,19,15,15,26,33,31,16,22,23,138,72 | 3 | 4 | 2 | 1 | 0 | 1 | 0 | 3 | 1 | 1 | 0 | 0 | 8 | 3
  Arthralgia 0,0,0,0,0,0,26,32,30,16,20,21,136,72 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 0 | 1 | 1 | 0 | 18 | 7
  Fatigue 0,0,0,0,0,0,26,32,30,16,20,21,137,72 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 4 | 2 | 0 | 0 | 23 | 14
  Headache0,0,0,0,0,0,26,32,30,16,20,21,138,72 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 8 | 3 | 2 | 1 | 29 | 19
  Loss appetite 0,0,0,0,0,0,26,32,31,16,22,23,138,72 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 8 | 5 | 2 | 2 | 2 | 20 | 12
  Myalgia0,0,0,0,0,0,26,32,30,16,20,21,138,72 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 5 | 2 | 1 | 0 | 29 | 11
  Nausea 0,0,0,0,0,0,26,32,30,16,20,21,137,72 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 2 | 0 | 0 | 17 | 10
  Body Temp. ( >= 38C ) | 4 | 8 | 2 | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 4 | 3
  Treatment of pain and or fever | 6 | 9 | 3 | 3 | 0 | 1 | 0 | 4 | 4 | 0 | 2 | 0 | 9 | 6

3. Primary Outcome: Number of Subjects Reporting Unsolicited Adverse Events Following Vaccination With Either TIVc or TIV by Overall Age Group and Age Sub-strata
Description: Safety was assessed in terms of number of subjects who reported any unsolicited AEs (four weeks after 1st vaccination and up to three weeks after 2nd vaccination), serious adverse events (SAEs), new onset of chronic diseases (NOCD), medically attended AEs and AEs leading to vaccine/study withdrawal after receiving one or two doses of either TIVc or TIV by overall age group (3 to <18 years) and age sub-strata (3 to <9 years and 9 to <18 years)
Time Frame: Day 1 -Day 181(one dose group) Day 1 -Day 209(two dose group)
Population: Analysis was done on unsolicited safety dataset, i.e. all subjects in the Exposed Set who have post-vaccination unsolicited AE records (even if no AEs have occurred)
Measure: Number; unit: Subjects
Groups:
- TIVc (3 to <18 Years): Vaccine naïve and non-naive subjects received one or two doses of cell culture derived trivalent subunit influenza vaccine formulation (TIVc)
- TIV (3 to <18 Years): Vaccine naïve and non-naive subjects received one or two doses of egg derived trivalent subunit influenza vaccine formulation (TIV)
- TIVc_Naive (3 to <9 Years): Vaccine naïve subjects received one dose of cell culture derived trivalent subunit influenza vaccine formulation (TIVc)
- TIVc_Non Naive (3 to <9 Years): Vaccine non naïve subjects received one dose of cell culture derived trivalent subunit influenza vaccine formulation (TIVc)
- TIV_Naive (3 to <9 Years): Vaccine naïve subjects received one dose of egg derived trivalent subunit influenza vaccine formulation (TIV)
- TIV_Non Naive (3 to <9 Years): Vaccine non naïve subjects received one dose of egg derived trivalent subunit influenza vaccine formulation (TIV)
Arm/Group | TIVc (3 to <18 Years) | TIV (3 to <18 Years) | TIVc_Naive (3 to <9 Years) | TIVc_Non Naive (3 to <9 Years) | TIVc_Non Naive (9 to <18 Years) | TIV_Naive (3 to <9 Years) | TIV_Non Naive (3 to <9 Years) | TIV_Non Naive (9 to <18 Years)
Number analyzed (Participants) | 278 | 148 | 85 | 54 | 139 | 39 | 35 | 74
Subjects
  Any AEs | 213 | 111 | 77 | 46 | 90 | 32 | 29 | 50
  Any possibly related AEs | 17 | 12 | 7 | 3 | 7 | 5 | 3 | 4
  SAEs | 12 | 4 | 4 | 2 | 6 | 0 | 2 | 2
  Possibly or probably related SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AEs leading to NOCD | 3 | 1 | 1 | 0 | 2 | 0 | 1 | 0
  Medically Attended AEs | 187 | 94 | 71 | 38 | 78 | 28 | 24 | 42
  AEs leading to vaccine/study withdrawal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local,systemic AEs collected -day 1 through Day 7 post injection 1 and Day 29 through Day 35 post injection 2, unsolicited AEs -Day 1 through Day 29 post 1st vaccination and Day 29 to Day 57 post 2nd vaccination. SAEs Day 1 through end of study
Description: Subjects 9 to <18 years of age were determined to be "previously vaccinated (vaccine non-naive)" by default. Analysis was done on unsolicited safety set-All subjects in the exposed set who had postvaccination unsolicited AE records (even if no AEs were reported).
Groups:
- Total: Total Number of subjects
Arm/Group | TIVc (3 to <18 Years) | TIV (3 to <18 Years) | Total
Serious Adverse Events (participants affected / at risk) | 12/278 | 4/148 | 16/426
Other Adverse Events (participants affected / at risk) | 246/278 | 126/148 | 372/426
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TIVc (3 to <18 Years) (N=278) | TIV (3 to <18 Years) (N=148) | Total (N=426)
LYMPHADENITIS (Blood and lymphatic system disorders) | 1 | 0 | 1
SICKLE CELL ANAEMIA WITH CRISIS (Blood and lymphatic system disorders) | 1 | 0 | 1
VOMITING (Gastrointestinal disorders) | 1 | 1 | 2
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 1 | 0 | 1
MASTOIDITIS (Infections and infestations) | 0 | 1 | 1
PHARYNGOTONSILLITIS (Infections and infestations) | 1 | 0 | 1
PNEUMONIA (Infections and infestations) | 2 | 0 | 2
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 1 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 1
COMPLEX PARTIAL SEIZURES (Nervous system disorders) | 1 | 0 | 1
HEADACHE (Nervous system disorders) | 1 | 0 | 1
TOXIC ENCEPHALOPATHY (Nervous system disorders) | 1 | 0 | 1
ANXIETY DISORDER (Psychiatric disorders) | 1 | 0 | 1
ASTHMATIC CRISIS (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
BRONCHOPNEUMOPATHY (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
HYPERTENSION (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TIVc (3 to <18 Years) (N=278) | TIV (3 to <18 Years) (N=148) | Total (N=426)
DIARRHOEA (Gastrointestinal disorders) | 26 | 8 | 34
NAUSEA (Gastrointestinal disorders) | 23 | 13 | 36
VOMITING (Gastrointestinal disorders) | 27 | 16 | 43
CHILLS (General disorders) | 36 | 9 | 45
FATIGUE (General disorders) | 31 | 16 | 47
INJECTION SITE ERYTHEMA (General disorders) | 32 | 32 | 64
INJECTION SITE HAEMORRHAGE (General disorders) | 17 | 13 | 30
INJECTION SITE INDURATION (General disorders) | 35 | 31 | 66
INJECTION SITE PAIN (General disorders) | 147 | 86 | 233
PYREXIA (General disorders) | 37 | 21 | 58
BRONCHITIS (Infections and infestations) | 21 | 12 | 33
GASTROENTERITIS (Infections and infestations) | 19 | 10 | 29
NASOPHARYNGITIS (Infections and infestations) | 35 | 19 | 54
OTITIS MEDIA ACUTE (Infections and infestations) | 14 | 3 | 17
PHARYNGITIS (Infections and infestations) | 22 | 12 | 34
RESPIRATORY TRACT INFECTION (Infections and infestations) | 14 | 5 | 19
TONSILLITIS (Infections and infestations) | 16 | 6 | 22
VIRAL INFECTION (Infections and infestations) | 16 | 6 | 22
DECREASED APPETITE (Metabolism and nutrition disorders) | 33 | 17 | 50
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 27 | 11 | 38
MYALGIA (Musculoskeletal and connective tissue disorders) | 40 | 14 | 54
HEADACHE (Nervous system disorders) | 42 | 26 | 68
SOMNOLENCE (Nervous system disorders) | 14 | 5 | 19
EATING DISORDER (Psychiatric disorders) | 17 | 7 | 24
IRRITABILITY (Psychiatric disorders) | 17 | 8 | 25
ASTHMATIC CRISIS (Respiratory, thoracic and mediastinal disorders) | 18 | 12 | 30
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 13 | 8 | 21
COUGH (Respiratory, thoracic and mediastinal disorders) | 26 | 10 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.